CLINICAL TRIAL: NCT03943251
Title: Safety, Tolerability, and Pharmacokinetics Phase ⅠStudy of a Selective Serotonin Partial Agonist and Reuptake Inhibitors, HEC113995PA•H2O, Following Single Ascending Doses，Single-center, Randomized, Double-blind in Healthy Subjects
Brief Title: The Study of a Selective Serotonin Partial Agonist and Reuptake Inhibitors, HEC113995PA•H2O,in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HEC113995PA•H2O-P-01/CRC-C19
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEC113995PA•H2O tablet (Experimental): Including 7 dose groups(2.5-、5、10-、20-、40-、60-、80mg).Each dose group was given only once.After an overnight stay of at least 10h on an empty stomach, 240mL of water was administered in the morning under the condition of an empty stomach. Water was forbidden for 1h before and 1h after administration, and fasting for 4h after administration.
  Interventions: Drug: HEC113995PA•H2O tablet
- placebo tablet (Placebo Comparator): Including 7 dose groups(2.5-、5、10-、20-、40-、60-、80mg).Each dose group was given only once.After an overnight stay of at least 10h on an empty stomach, 240mL of water was administered in the morning under the condition of an empty stomach. Water was forbidden for 1h before and 1h after administration, and fasting for 4h after administration.
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: HEC113995PA•H2O tablet — 2.5-、5-、10-、20-、40-、60-、80mg HEC113995PA•H2O tablet in day1.
  Arms: HEC113995PA•H2O tablet
Drug: Placebo tablet — 2.5-、5-、10-、20-、40-、60-、80mg Placebo tablet in day1.
  Arms: placebo tablet

SUMMARY:
This study is a safety, tolerability, and pharmacokinetics phase Ⅰstudy of a selective Serotonin partial agonist and reuptake inhibitors, HEC113995PA•H2O,in healthy subjects.This study is the healthy adult subjects single ascending-dose research.

DETAILED DESCRIPTION:
There have set up seven dose group(2.5、5、10、20、40、60、80mg）.The first group(2.5mg)contains 8 health subjects(6 health subjects take experimental drugs,2 health subjects take the placebo). Other groups contains 10 health subjects(8 health subjects take experimental drugs,2 health subjects take the placebo).Within 30min before taking the medicine and after 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 10h, 24h, 36h, 48h,72h to take blood samples for pharmacokinetics(PK) detection.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study, able to understand and sign the informed consent, and able to complete the the study in accordance with the requirements of the study.
* Female subjects who are not pregnant or lactating and male subjects whose female partners are fertile shall voluntarily take effective contraceptive measures from the date of signing the informed consent form to 3 months after the medication.
* When signing the informed consent, 18 years old ≤the age≤45 years old, gender is not limited.
* Male body weight ≥50kg, female body weight ≤45kg, and body mass index (BMI) in the range of 18-28 kg/m2 (including the critical value).
* No clinical significance of vital signs, physical examination, laboratory examination, chest X-ray (posterior and anterior) and electrocardiogram results.

Exclusion Criteria:

* The serum creatinine, ALT and AST levels ≥1.5 times of the normal upper limit in the screening period.
* The HbsAg, anti-HCV, HIV-antibody or syphilis antibody is positive in screening.
* Patients with clinical significance of the following diseases, including but not limited to gastrointestinal, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular diseases, epilepsy, bipolar disorder/mania, high intraocular pressure or acute angle-closure glaucoma disease history.
* Those who are known to have allergy history or allergy constitution to the test preparation and any of its components or related preparations.
* Any prescription or over-the-counter medication taken within 14 days prior to starting the study drug, or any drug that inhibits or induces the liver to metabolize the drug within 28 days [e.g., inducer - the barbiturates, rifampicin, carbamazepine, phenytoin, omeprazole, griseofulvin, ammonia methyl propyl ester, etc.; inhibitors - large ring lactone class antibiotic (such as erythromycin, clarithromycin, etc.), azole antifungal drugs (such as ketone health zun, itraconazole, etc.), fluoroquinolone (e.g., ciprofloxacin, sand magnitude), calcium channel blockers (such as verapamil, diltiazem, etc.), H1 receptor antagonist (e.g., astemizole, etc.), H2 receptor antagonist (e.g., cimetidine, etc.), SSRI antidepressants (such as fluoxetine, fluvoxamine, etc.), benzodiazepines a tranquilizer, clopidogrel, gemfibrozil, deferasirox, teriflunomide, telithromycin, trimethoprim, HMG-CoA reductase inhibitors (such as lovastatin, simvastatin, etc.), nitroimidazoles, etc.
* Those who ingested food or drink containing caffeine, xanthine, alcohol or grapefruit within 48 hours before taking the study drug.
* The urine drug abuse screening(morphine, tetrahydrocannabinolate, methamphetamine, dimethylene dioxyamphetamine, ketamine, and cocaine) is positive.
* Intemperant or regular drinkers within 3 months prior to the study, i.e., those who consumed more than 21 units of alcohol per week (1 unit =360mL beer or 45mL spirit with 40% alcohol or 150mL wine), or those who were positive on the alcohol breath test.
* A heavy smoker or smokers who smoke more than 10 cigarettes per day within 3 months prior to administration or who fail to comply with the no smoking regulation during the study.
* Those who had a blood donation or blood loss of >400mL within one month before taking the study drug.
* Those who plan to receive an organ transplant or have had one.
* Those who have participated in clinical trials of other drugs within 3 months before randomization.
* Subjects considered by the investigator to have other factors unsuitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Adverse events of the single ascending-dose | From the baseline to day4
  To assess the safe and tolerability of the single ascending-dose

SECONDARY OUTCOMES:
Maximum Plasma Concentration(Cmax) | Prior to dosing（0.5h）and 0.5h,1h,1.5h,2h,2.5h,3h,4h,5h,6h,8h,10h,12h,24h,36h,48h,72h after dosing
  Maximum Plasma Concentration(Cmax)of HEC113995PA•H2O in single ascending-dose
Area Under the Curve(AUC) | Prior to dosing（0.5h）and 0.5h,1h,1.5h,2h,2.5h,3h,4h,5h,6h,8h,10h,12h,24h,36h,48h,72h after dosing
  Area Under the Curve(AUC) of HEC113995PA•H2O in single ascending-dose
Maximum Peak Time(Tmax) | Prior to dosing（0.5h）and 0.5h,1h,1.5h,2h,2.5h,3h,4h,5h,6h,8h,10h,12h,24h,36h,48h,72h after dosing
  Maximum Peak Time(Tmax) of HEC113995PA•H2O in single ascending-dose

OTHER OUTCOMES:
Mean Residence Time(MRT) | Prior to dosing（0.5h）and 0.5h,1h,1.5h,2h,2.5h,3h,4h,5h,6h,8h,10h,12h,24h,36h,48h,72h after dosing
  Mean Residence Time(MRT) of HEC113995PA•H2O in single ascending-dose
Terminal elimination half-life(T1/2) | Prior to dosing（0.5h）and 0.5h,1h,1.5h,2h,2.5h,3h,4h,5h,6h,8h,10h,12h,24h,36h,48h,72h after dosing
  Terminal elimination half-life(T1/2) of HEC113995PA•H2O in single ascending-dose

CONTACTS AND LOCATIONS:
Locations (1):
- The Shanghai xuhui district central hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No